CLINICAL TRIAL: NCT05385536
Title: Evaluating UTI Outcomes in at Risk Populations
Acronym: At Risk
Status: Completed | Type: Observational
Sponsor: Pathnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-PARS
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Urinary Tract Infections; Complicated Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Guidance clinical pathway: Sites will be provided a standardized infrastructure and process for collecting and reporting of urine test results including unique lab requisitions that contain the option to order Guidance® UTI, Standard Urine Culture (SUC), and Urine Analysis (UA) along with a protocol for results notification.
- Traditional clinical pathway: Sites will employ their current standard clinical care practices for suspected UTI, including Standard Urine Culture (SUC), Urine Analysis (UA), and Guidance® UTI testing as per current reporting practices. Providers at these facilities will have the option to order any diagnostic test they deem appropriate.

SUMMARY:
This is a multicenter, observational comparative cohort, study to evaluate the UTI related adverse event rates between Guidance® UTI clinical pathway versus the current traditional clinical pathways for urine testing.

DETAILED DESCRIPTION:
Clinical sites will be identified by an internal database, prepared by the sponsor, based on previous experience with the sites. Study allocation will based on their current usage of Guidance® UTI and the reporting pathway (described above) will be implemented. Those who currently routinely use Guidance® UTI testing procedures will be over sampled 2:1 over those who do not routinely use Guidance® UTI. Larger clinical care systems with multiple care sites may have locations allocated to different cohort. The basis for cohort allocation will be based on the availability and willingness of providers in these markets to implement infrastructure for collecting and reporting of Guidance® UTI clinical pathway. The comparative cluster cohort will be selected from select geographies within the U.S. based on size of general population served matching to those enrolled in the Guidance® UTI clinical pathway.

The method of patient care and management (e.g., test ordering and antimicrobial initiation) is at the discretion of the treating physicians. Specimens collected for suspected UTI may be sent to Pathnostics for standard bacterial identification and sensitivities. Guidance® UTI can only be performed at Pathnostics, whereas urine cultures may be performed at any lab. Trained and experienced clinical lab scientists at Pathnostics are always available to assist the ordering provider with results interpretation or any other questions on the report they may have.

ELIGIBILITY:
Inclusion

* Male or female participants ≥ 65 years of age, no predetermined quotas or ratios for gender participation.
* High suspicion of active UTI
* Ability to provide/obtain a clean catch or sterile urine specimen
* Willing to adhere to follow-up schedule as stated in schedule of events
* Permanent residence in the same state in which they were consented for the study
* Able to provide informed consent

Exclusion

* Participation in another UTI trial during the study period
* Patients in hospice-care or limited life expectancy of ≤1 month)
* Inability to provide informed consent and/or respond independently to follow up surveys
* If the provider deems that a urine culture or Guidance UTI is not necessary in clinical management

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 65 years of age seen by healthcare professional for UTI
Sampling Method: Non-Probability Sample
Enrollment: 7921 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
UTI-related ED visit and/or hospitalization within 30 days of index visit | within 30 days of index visit
  UTI-related ED visit and/or hospitalization within 30 days of index visit
Composite of adverse events associated with index UTI event | within 30 days of index visit
  Composite of adverse events associated with index UTI event
  Allergic reactions to antibiotic therapy
  Progression to pyelonephritis
  Nausea/vomiting, headache, skin rash, anaphylaxis/hypersensitivity reaction
  yeast infection (Vaginitis/vulvovaginal candidiasis)
  Progression to acute renal failure
  Tendinopathy (including tendon rupture)
  C. difficile infection
  Sepsis
Recurrent UTI (rUTI) - The proportion of subjects reporting recurrence of symptomatic UTI and receive antimicrobial treatment (re-prescription) within 30 days. | within 30 days of index visit
  Recurrent UTI (rUTI) - The proportion of subjects reporting recurrence of symptomatic UTI and receive antimicrobial treatment (re-prescription) within 30 days.

SECONDARY OUTCOMES:
Rate of empirical antibiotic starts for UTI indication | within 1 year of index visit
  Rate of empirical antibiotic starts for UTI indication
Rate of antimicrobial changes for UTI indication | within 1 year of index visit
  Rate of antimicrobial changes for UTI indication
Recurrent UTI within 1 year of index visit suspected UTI as measured by total antibiotics prescribed. | within 1 year of index visit
  Recurrent UTI within 1 year of index visit suspected UTI as measured by total antibiotics prescribed.
UTI-related ED visit and/or hospitalization within 1 year of index visit | within 1 year of index visit
  UTI-related ED visit and/or hospitalization within 1 year of index visit

CONTACTS AND LOCATIONS:
Locations (1):
- Dispatch Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No